CLINICAL TRIAL: NCT03121079
Title: Interferon-α Prevents Leukemia Relapse of AML Patients Undergoing HLA-identical Allogeneic Hematopoietic Stem Cell Transplantation With Pretransplant MRD
Brief Title: Interferon-α Prevents Leukemia Relapse of AML Patients After Transplantation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: there was almost no patient would enroll in this study.
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaojun Huang,MD, Director of Peking University Institute of Hematology, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017PHB013-01
Record Dates: First submitted 2017-04-14; First posted 2017-04-19 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Interferon-A-2B; Relapse; Prevention; Hematopietic Stem Cell Transplantation
Keywords: Interferon-alpha; Relapse; prevention; hematopietic stem cell transplantation; acute myeloid leukemia
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute | interventions — Interferon-alpha

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interferon alpha group (Experimental): The patients in arm will be receive interferon alpha injection (3 million U/time)twice a week, as the intervention since the third month after HLA-identical transplantation.
  Interventions: Drug: Interferon-alpha

INTERVENTIONS:
Drug: Interferon-alpha — patients in Interferon-alpha group will receive Interferon-alpha injection since the third month after transplantation for six months.

SUMMARY:
Allogeneic stem cell transplantation (SCT) remains a powerful therapeutic modality for patients with acute myeloid leukemia (AML).The superior clinical outcomes of allogeneic human SCT versus chemotherapy alone as post-remission treatment could be related to the graft-versus-leukemia (GVL) effects of recovered donor T cells. Our previous study investigated both the association of MRD status with transplant outcomes in haplo-SCT and matched sibling donor transplantation(MSDT)， and also possible differences in the transplant outcomes of patients with positive pre-MRD (as determined by MFC) who underwent haplo-SCT versus MSDT. It provided new evidence that unmanipulated haplo-SCT is superior to matched sibling donor transplantation in eradicating pre-transplantation MRD, indicating that unmanipulated haploidentical allografts have stronger GVL effects.As to the AML patients in standard-risk, who have a positive MRD before MSDT, whether these patients should be given any relapse prevention is the question to be answered in this study. Interferon α-2b exerts a relatively strong immunomodulatory effect. It can kill AL cells by regulating T-cell and/or natural killer cell functions.Consequently, interferon α-2b may have potential value for high-risk AL patients after transplantation. The study hypothesis: Using interferon α-2b following hematopoietic stem cell transplantation in patients with standard-risk AML can further reduce relapse rate and improve leukemia-free survival.

DETAILED DESCRIPTION:
The standard-risk AML patients (18-60 years) receiving HLA-identical allogeneic stem cell transplantation in Peking University Institute of Hematology will be enrolled in this study if their MRD were positive before SCT, in CR1/CR2, remain in CR and MRD negative in the first two months after transplantation. The patients in this study will be treated with interferon-alpha injection twice a week (3 million units / time, iH) since the third month posttransplant. If the patients were well tolerated, the interferon-alpha treatment will continue 6 months. All the enrolled patients will undergo MRD monitoring after SCT as the same as the routine procedure. Bone marrow examination will be performed at the regular time points (+1, 2,3, 4, 5, 6, 9, 12 month) and 8-colour flow cytometry and RQ-PCR-based WT1 examination will be empolyed to evaluate MRD and disease status. Based on the statistical calculation, in order to reduce the incidence of relapse from 40% (previous data) to 15% (the cumulative incidence of relapse in pre-MRD- AML patients), total 29 patients will be enrolled. The main side effects might related to interferon-alpha include induction of severe GVHD, hematological toxicity and Flu - like symptoms. If the patients met the following criteria, they will withdraw from the trial: 1）met the combined criteria for positive MRD (MRDco+) which was defined as 2 consecutive FCM+ or WT1+ results or both FCM+ and WT1+ in a single sample within 1 year after transplantation; 2）hematological relapse; 3) grade III or IV acute GVHD, or moderate/ severe chronic GVHD; 4) severe infection; 5) grade IV hematological toxicity; 6) organ failure; 7) death; 8) patients refuse to continue the interferon-alpha treatment. The main end point of the study is one-year cumulative incidence of relapse. the second end points include OS, NRM, DFS, MRD, GVHD, infection and hematological toxicity.

ELIGIBILITY:
Inclusion Criteria:

* standard-risk AML in CR1/CR2
* without t(9;22) and t(15;17)
* receive HLA-identical transplantation
* with positive MRD before transplantation (measured by flow cytometry)
* CR within the first two months posttransplantation and MRD is negative
* between 18-60 years

Exclusion Criteria:

* uncontrolled GVHD
* be in myelosuppression (WBC<1.5x10^9/L, ANC<0.5×10^9/L，PLT<25×10^9/L,HB<65g/L)
* severe infection
* organ failure
* the patients do not agree to participate in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
cumulative incidence of relapse | within the first year after transplantation
  the cumulative incidence of relapse

SECONDARY OUTCOMES:
OS | within the first year after transplantation
  overall survival
NRM | within the first year after transplantation
  non-relapse motality
DFS | within the first year after transplantation
  disease-free survival
MRD | within the first year after transplantation
  cumulative incidence of MRD+
acute GVHD | within 100 days after transplantation
  acute graft-versus-host disease
chronic GVHD | within the first year after transplantation
  chronic graft-versus-host disease
infection | within the first year after transplantation
  bacteria, fungal, virus, etc.

OTHER OUTCOMES:
Hematologic toxicity | within the first year after transplantation
  any decrease of blood cells including white, red blood cells and platelet

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Huang, Dr., Principal Investigator — Peking University Institute of Hematology
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No